CLINICAL TRIAL: NCT03274440
Title: Effects of Marijuana on Symptoms of Obsessive-Compulsive Disorder
Brief Title: Effects of Marijuana on Symptoms of OCD
Acronym: ECOS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Reilly R. Kayser, Resident, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: # 7405
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Marijuana; THC; Cannabis; CBD; Cannabinoid
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High THC/Low CBD Marijuana (Experimental): This condition involves the ingestion of marijuana with a high THC (5-10%) and low CBD (<1%) content.
  Interventions: Drug: Cannabis
- Low THC/High CBD Marijuana (Experimental): This condition involves the ingestion of marijuana with a low THC (<1%) and high CBD (>10%) content.
  Interventions: Drug: Cannabis
- No THC/No CBD (Placebo Comparator): This condition involves the ingestion of a placebo control with no THC and no CBD content.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabis — THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
  Other Names: marijuana
  Arms: High THC/Low CBD Marijuana; Low THC/High CBD Marijuana
Other: Placebo — Placebo control group, not receiving THC or CBD.
  Arms: No THC/No CBD

SUMMARY:
The purpose of this pilot research study is to test whether certain components of the marijuana plant, known as "cannabinoids", may help to reduce symptoms in patients with OCD. Specifically, patients enrolled in the study will smoke marijuana containing different concentrations of 2 different cannabinoids, THC and CBD. Both of these agents act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD. Neither compound is currently FDA-approved for treating OCD.

DETAILED DESCRIPTION:
Prior research suggests that certain areas of the brain are receptive to chemicals like those found in the cannabis (marijuana) plant, known as cannabinoids, and that these regions may be involved in anxiety disorders and OCD. More recent data shows that synthetic drugs that target these systems may be helpful in conditions related to OCD like anxiety disorders and Tourette's syndrome. Thus, these substances could also possibly be useful to treat OCD symptoms. However, to date there has been little research regarding the role of cannabinoids in OCD.

The purpose of this study is to examine the effects of different cannabinoids on OCD symptoms in humans. To accomplish this in a laboratory setting, patients with OCD who are also occasional cannabis users will receive different combinations of two of the most well-studied cannabinoids, delta-9-tetrahydrocannabinol (THC, the main psychoactive component in cannabis) and cannabidiol (CBD, another component of the cannabis plant). We will then measure acute effects on OCD symptoms, anxiety, intoxication, and cardiovascular outcomes (i.e. blood pressure and heart rate).

ELIGIBILITY:
Inclusion Criteria:

* Age 21-55
* Physically healthy
* Diagnosed with OCD
* Current marijuana user
* Women of childbearing potential must be using an effective form of birth control
* Not currently taking psychotropic medications
* Ability to provide informed consent

Exclusion Criteria:

* History of any significant medical condition that may increase the risk of participation
* Females who are pregnant or nursing
* If female, not pregnant
* Current or lifetime history of psychiatric disorders other than OCD that may increase the risk of participation
* Current substance use disorder
* Severe depression or positive urine toxicology (other than THC) at screening, or any adverse reaction to a cannabinoid
* Patients who are seeking treatment for substance abuse
* Patients who are planning to begin a course of cognitive-behavioral therapy within 8 weeks of beginning the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reilly Kayser, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to receive high THC/low CBD cannabis ("THC"), low THC/high CBD cannabis ("CBD"), and placebo cannabis ("PBO"). Total participants for each order were:
  Order A (THC, CBD, PBO) = 3 Order B (THC, PBO, CBD) = 2 Order C (CBD, THC, PBO) = 4 Order D (CBD, PBO, THC) = 1 Order E (PBO, THC, CBD) = 1 Order F (PBO, CBD, THC) = 3
Pre-assignment Details: Participants who met study criteria and chose to participate were assigned to receive each of the three study conditions (high THC/low CBD; low THC/high CBD; placebo with no THC or CBD) in random order. All sessions were separated by at least 1 calendar week.
Groups:
- Order A: Order A: THC, CBD, PBO.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
- Order B: Order B: THC, PBO, CBD.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
- Order C: Order C: CBD, THC, PBO.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
- Order D: Order D: CBD, PBO, THC.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
- Order E: Order E: PBO, THC, CBD.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
- Order F: Order F: PBO, CBD, THC.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
Period: Overall Study
Arm/Group | Order A | Order B | Order C | Order D | Order E | Order F
Started | 3 | 2 | 4 | 1 | 1 | 3
Completed | 2 | 2 | 4 | 0 | 1 | 3
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Time commitment too great | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for all study completers
Groups:
- All Participants: In this within-subjects study, all participants received all three study drugs in random order. Demographic data is provided for all study participants together.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Psychiatric Comorbidity [Count of Participants; unit: Participants] — Comorbid psychiatric conditions (other than OCD)
  Participants
    Major Depressive Disorder (MDD) | 2
    Generalized Anxiety Disorder (GAD) | 2
    Panic Disorder | 1
    None | 8
Medication Status [Count of Participants; unit: Participants] — Number of patients taking psychotropic medication
  Participants
    Selective Serotonin Reuptake Inhibitor (SSRI) | 2
    Unmedicated | 10
Cannabis use at time of enrollment [Mean (Standard Deviation); unit: days per week] — Self-reported cannabis use (number of days per week) at time of enrollment
  days per week | 3.8 (2.9)
Yale-Brown Obsessive-Compulsive Scale (YBOCS) [Mean (Standard Deviation); unit: units on a scale] — A scale measuring OCD symptom severity. Total score is reported and ranges from 0 (no symptoms) to 40 (severe symptoms). Scores >16 are consistent with clinical OCD symptoms.
  units on a scale | 20.1 (4.9)
Speilberger State-Trait Anxiety Scale, Trait Version (STAI-T) [Mean (Standard Deviation); unit: units on a scale] — A scale measuring trait anxiety. Total score is reported and ranges from 20 (no trait anxiety) to 80 (severe trait anxiety). The norm for adults is 34.9+/-9.2.
  units on a scale | 48.5 (13.9)
Hamilton Depression Rating Scale, 17-Item (HDRS-17) [Mean (Standard Deviation); unit: units on a scale] — A scale measuring depression symptoms. Total score is reported and ranges from 0 (no depression) to 52 (most severe depression).
  Anchors:
  0-7 = no depression 8-16 = mild depression 17-25 = moderate depression >25 = severe depression
  units on a scale | 4.9 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive-Compulsive Challenge Scale (YBOC-CS)
Description: An adapted version of the Yale-Brown Obsessive-Compulsive Scale (YBOCS) which measures change in OCD symptoms over short time frames (i.e., since the last assessment as opposed to over the past week). Total score is reported. Scores range from 0 (no symptoms) to 40 (severe symptoms).
Time Frame: Baseline was obtained at the beginning of each session. Then, change from baseline was measured following cannabis administration (minute 0) at minutes 20, 40, 60, 90, 120, and 180. This procedure was repeated for each of the 3 conditions.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High THC/Low CBD Marijuana (Cannabis): This condition involves the ingestion of marijuana (cannabis) with a high THC (5-10%) and low CBD (<1%) content.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
- Low THC/High CBD Marijuana (Cannabis): This condition involves the ingestion of marijuana (cannabis) with a low THC (<1%) and high CBD (>10%) content.
  Cannabis: THC and CBD are "cannabinoids" which are found naturally in the marijuana plant. Both act on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
Arm/Group | High THC/Low CBD Marijuana (Cannabis) | Low THC/High CBD Marijuana (Cannabis) | No THC/No CBD
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Minute 0 (baseline) | 17.45 (7.46) | 17.00 (8.07) | 17.09 (4.16)
  Minute 20 | 13.36 (10.15) | 11.55 (9.46) | 10.91 (3.70)
  Minute 40 | 11.09 (6.82) | 11.64 (9.91) | 9.00 (2.59)
  Minute 60 | 10.18 (5.90) | 11.18 (10.15) | 9.27 (3.69)
  Minute 90 | 9.00 (4.80) | 9.91 (7.62) | 12.18 (7.44)
  Minute 120 | 9.00 (5.44) | 9.64 (5.89) | 11.09 (6.80)
  Minute 180 | 10.18 (6.35) | 11.64 (10.12) | 10.00 (4.77)
Statistical Analysis 1: Comparison: High THC/Low CBD Marijuana (Cannabis) vs Low THC/High CBD Marijuana (Cannabis) vs No THC/No CBD; Test for interaction effect between condition and time (includes all three groups and all time points); Test type: Other — A random-effects linear mixed model evaluated changes in YBOCCS as a function of condition (THC, CBD, placebo [PBO]), time point, and their interaction; p = .577, Linear mixed effects regression
Statistical Analysis 2: Comparison: High THC/Low CBD Marijuana (Cannabis) vs Low THC/High CBD Marijuana (Cannabis) vs No THC/No CBD; Test for main effect of time (includes all three groups and all time points); Test type: Other — [test comment as in outcome 1, analysis 1]; p < .001, Linear mixed effects regression; F=10.50; df=6, 10
Statistical Analysis 3: Comparison: High THC/Low CBD Marijuana (Cannabis) vs Low THC/High CBD Marijuana (Cannabis) vs No THC/No CBD; Test for main effect of condition (includes all three groups and all time points); Test type: Other — [test comment as in outcome 1, analysis 1]; p = .72, Linear mixed effects regression

2. Secondary Outcome: Spielberger State-Trait Anxiety Scale: State Version (STAI-S)
Description: A scale measuring state (acute) anxiety. Total score is reported. Scores range from 20 (no state anxiety) to 80 (severe state anxiety).
Time Frame: Baseline obtained at the beginning of the session (Minutes 0), and then the scale was obtained at minutes 20, 40, 60, 90, 120, and 180 after cannabis administration.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High THC/Low CBD Marijuana (Cannabis) | Low THC/High CBD Marijuana (Cannabis) | No THC/No CBD
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Minute 0 (baseline) | 44.18 (15.37) | 45.00 (14.30) | 42.27 (10.87)
  Minute 20 | 40.00 (21.37) | 37.55 (15.28) | 29.73 (7.64)
  Minute 40 | 36.00 (13.54) | 36.00 (15.63) | 29.36 (7.37)
  Minute 60 | 33.00 (10.49) | 36.82 (14.83) | 32.27 (9.77)
  Minute 90 | 34.91 (11.48) | 34.64 (10.56) | 35.91 (10.17)
  Minute 120 | 35.09 (12.47) | 35.18 (8.67) | 34.09 (9.74)
  Minute 180 | 35.18 (10.65) | 37.45 (15.64) | 32.45 (9.27)
Statistical Analysis 1: Comparison: High THC/Low CBD Marijuana (Cannabis) vs Low THC/High CBD Marijuana (Cannabis) vs No THC/No CBD; Test for interaction between condition and time; Test type: Other — A random-effects linear mixed model evaluated changes in STAI-S as a function of condition (THC, CBD, placebo [PBO]), time point, and their interaction; p = .577, Linear mixed effects regression
Statistical Analysis 2: Comparison: High THC/Low CBD Marijuana (Cannabis) vs Low THC/High CBD Marijuana (Cannabis) vs No THC/No CBD; Test for main effect of time; Test type: Other — [test comment as in outcome 2, analysis 1]; p < .001, Linear mixed effects regression; F=7.00, df=6,10
Statistical Analysis 3: Comparison: High THC/Low CBD Marijuana (Cannabis) vs Low THC/High CBD Marijuana (Cannabis) vs No THC/No CBD; Test for main effect of condition; Test type: Other — [test comment as in outcome 2, analysis 1]; p = .002, Linear mixed effects regression; F=6.26, df=2, 10

ADVERSE EVENTS:
Time Frame: Over the course of all 3 sessions, an average of 38 days.
Description: Participants in this preliminary study were randomized to receive high THC/low CBD cannabis ("THC"), low THC/high CBD cannabis ("CBD"), and inert placebo cannabis ("PBO"), in random order. The total number of participants who received each possible order is listed below:
  Order A (THC, CBD, PBO) = 2 Order B (THC, PBO, CBD) = 2 Order C (CBD, THC, PBO) = 4 Order D (CBD, PBO, THC) = 0 Order E (PBO, THC, CBD) = 1 Order F (PBO, CBD, THC) = 3
Groups:
- High THC/Low CBD Cannabis: Adverse events after receiving High THC (5-10%)/Low CBD (<1%) cannabis
- High CBD/Low THC Cannabis: Adverse events after receiving Low THC (<1%)/High CBD (5-10%) cannabis
- Placebo Cannabis: Adverse events after receiving placebo (0% THC/ 0% CBD) cannabis
Arm/Group | High THC/Low CBD Cannabis | High CBD/Low THC Cannabis | Placebo Cannabis
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03274440/Prot_SAP_ICF_000.pdf